CLINICAL TRIAL: NCT03500536
Title: Implementing an Innovative Suite of Mobile Applications for Depression and Anxiety
Brief Title: Understanding the Efficacy of Mobile Apps as Intervention for Depression in Adults When Deployed as Part of Primary Care.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Actualize Therapy (Industry)
Collaborators: University of Arkansas (Other)
Responsible Party: Principal Investigator, Pauli Lieponis, Interim Principal Investigator, Actualize Therapy
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Main
Record Dates: First submitted 2018-04-10; First posted 2018-04-18 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Depression; Anxiety; Primary Health Care
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Waitlist Control (No Intervention): 8 weeks of treatment as usual followed by 8 weeks of IntelliCare treatment.
- Experimental (Experimental): 8 weeks of IntelliCare treatment followed by 8 weeks of treatment as usual.
  Interventions: Behavioral: IntelliCare

INTERVENTIONS:
Behavioral: IntelliCare — A suite of mobile apps that use principles of computerized therapy to decrease symptoms of depression.
  Arms: Experimental

SUMMARY:
The clinical study is meant to optimize the mobile intervention, to develop a robust implementation plan for the mobile intervention within primary care, and to conduct an effectiveness trial, randomizing 128 participants in order to understand effect on severity of depression and anxiety symptoms, cost-effectiveness, and usability of mobile apps.

ELIGIBILITY:
Inclusion Criteria:

* Positive screen on PHQ-9

Exclusion Criteria:

* Does not own or use a mobile smart phone

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2019-04-04 (Actual); Study Completion 2019-04-04 (Actual)

PRIMARY OUTCOMES:
Symptoms of depression | 8 weeks
  Using the PHQ-9 screener

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Graham AK, Greene CJ, Kwasny MJ, Kaiser SM, Lieponis P, Powell T, Mohr DC. Coached Mobile App Platform for the Treatment of Depression and Anxiety Among Primary Care Patients: A Randomized Clinical Trial. JAMA Psychiatry. 2020 Sep 1;77(9):906-914. doi: 10.1001/jamapsychiatry.2020.1011. PMID 32432695